CLINICAL TRIAL: NCT05928754
Title: Prospective CoHoRt Of Non-infectious Intermediate, pOsterior or panuveitiS
Acronym: CHRONOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P22-01
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Non-infectious Uveitis
Keywords: non-infectious uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uveitis Patients (Experimental): Uveitis Patients: intermediate, posterior or panuveitis noninfectious uveitis with Inflammatory activity requiring treatment with either one or more of the following:
  1. Systemic corticosteroids or periocular or intravitreal injections of corticosteroids
  2. Immunosuppressants: methotrexate, azathioprine, ciclosporine….
  3. Biotherapy: infliximab, adalimumab, tocilizumab
  Interventions: Diagnostic Test: care strategy
- Control Patients (Active Comparator): scheduled for cataract or vitreoretinal surgery
  Interventions: Diagnostic Test: care strategy

INTERVENTIONS:
Diagnostic Test: care strategy — Uveitis patients:
  * Blood sample (20ml): Additional 20 ml blood sample during the first visit and potentially during follow-up (if necessary) for the purpose of the biological collection;
  * Ocular sample (aqueous humor, vitreous): if required by the clinical context for the needs of the biological collection;
  * Specific imaging: adaptive optics or Doppler holography, these procedures will be indicated on a case-by-case basis, at the investigator's discretion, and concern only patients with inflammatory vascular damage (5 to 10% of patients in the uveitis cohort);
  * Quality of Life NEI-VFQ 25: provided at the inclusion visit and at follow-up visits M3-V2, M12-V5 and M24-V7.

SUMMARY:
prospective, cohort, longitudinal, multicenter, non-randomized study of patients with non-infectious posterior segment uveitis or panuveitis, with a group of control patients (scheduled for cataract or vitreoretinal surgery) and constitution of biological collection.

DETAILED DESCRIPTION:
Description of the clinical characteristics and evolution in a large cohort of patients with non-infectious uveitis, allowing to identify prognostic or predictive factors of response after treatment of these different forms of non-infectious uveitis of the posterior segment or panuveitis (factors that are currently not well known).

Uveitis patients:

* Blood sample (20ml): Additional 20 ml blood sample during the first visit and potentially during follow-up (if necessary) for the purpose of the biological collection;
* Ocular sample (aqueous humor, vitreous): if required by the clinical context for the needs of the biological collection;
* Specific imaging: adaptive optics or Doppler holography, these procedures will be indicated on a case-by-case basis, at the investigator's discretion, and concern only patients with inflammatory vascular damage (5 to 10% of patients in the uveitis cohort);
* Quality of Life NEI-VFQ 25: provided at the inclusion visit and at follow-up visits M3-V2, M12-V5 and M24-V7.

Control patients:

* Blood sample (20ml): Additional 20 ml blood sample during the inclusion visit at the time of the surgical scheduled procedure for the needs of the biological collection;
* Ocular sample (aqueous humor, vitreous): considered as surgical waste, the tissue residues will be collected during the scheduled surgical procedure for cataract or vitreoretinal surgery for the needs of the biological collection;

ELIGIBILITY:
Inclusion Criteria:

UVEITIS Patients:

* Adult patients (≥ 18 years);
* Non-infectious uveitis;
* Intermediate, posterior or panuveitis;
* Inflammatory activity requiring treatment with either one or more of the followings:

  * Systemic corticosteroids or periocular or intravitreal injections of corticosteroids;
  * Immunosuppressants: methotrexate, azathioprine, cyclosporine, etc.;
  * Biotherapy: infliximab, adalimumab, tocilizumab;
* Patients with health insurance;
* Written Informed consent obtained at enrolment in the study.

Control patients:

* Adult patients (≥ 18 years);
* Scheduled patients ( Non-urgente procedure) for cataract or vitreoretinal surgery;
* Patients with health insurance;
* Written Informed consent obtained at enrolment in the study.

Exclusion Criteria:

Uveitis Patients:

* Isolated anterior uveitis ;
* Inactive disease defined as:

  * Absence of inflammatory chorioretinal and/or inflammatory retinal vascular lesion;
  * Anterior chamber cell grade< 0.5+;
  * Vitreous haze grade <0.5+;
* Pregnant or breastfeeding woman at the inclusion visit;
* Patient under legal protection (" curatelle " or " tutelle ");
* Patient denied freedom by a legal or administrative order.

Control patients:

* Pregnant or breastfeeding woman;
* Unscheduled (urgent) cataract or vitreoretinal surgery;
* Patient under legal protection (" curatelle " or " tutelle ");
* Patient denied freedom by a legal or administrative order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Imaging database development | 60 months
  To develop an imaging database of Non-Infectious Uveitis of the posterior segment (NIUPS) using multimodal imaging
Biological constitution | 60 months
  To Constitute a biological collection of ocular and blood samples of NIUPS patients and controls
medico economic costs estimation | 60 months
  To estimate the current costs of treatment by ensuring linkage of cohort patients to the national claims database

IPD SHARING:
Plan to Share IPD: No